CLINICAL TRIAL: NCT04417244
Title: Complications of Adenovirus Keratoconjunctivitis in Ophthalmologists and Orthoptists: Epidemiology and Risk Factor, a Retrospective Questionnaire Analysis
Brief Title: Adenovirus Keratoconjunctivitis and Ophtalmology
Acronym: ADV-OPH
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Other Study IDs: 2020 ADV-OPH
Record Dates: First submitted 2020-06-02; First posted 2020-06-04 (Actual); Last update posted 2020-06-04 (Actual); Status verified 2020-05

CONDITIONS: Adenoviral Keratoconjunctivitis
Keywords: Adenovirus; Epidemic Keratoconjunctivitis; Subepithelial infiltrates; Occupational diseases; Ophtalmologists; Orthoptists; Epidemiology
MeSH Terms: conditions — Adenoviridae Infections; Occupational Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Adenovirus conjunctivitis is an epidemic disease registered as a common occupational disease for ophthalmologists and orthoptists. It can leave corneal sequelae even several years after infection.

The primary aim of the study is to investigate the prevalence of these sequelae in the at-risk population of ophthalmologists and orthoptist.

Secondary aim are to describe administrative procedures (occupational disease declaration and sick leave),infections characteristics; and risk factors.

DETAILED DESCRIPTION:
Adenovirus conjunctivitis is an epidemic disease registered as a common occupational disease for ophthalmologists and orthoptists. It can leave corneal sequelae even several years after infection.

The investigation tream create a nationwide anonymous retrospective questionnaire using the secure internet application REDCap® to build and manage the questionnaire addressed to ophtalmologists (interns, graduates and retirees) and orthoptists.

Investigator collect several characteristics such as general characteristics (sex, age range, profession), administrative procedure declaration (occupational disease declaration, sick leave, cessation of surgery); infection characteristics (bilaterality, season, anteriority, sequels, current therapy, professional discomfort), risk factor (refractive surgery history, wearing of eyeglasses or contact lenses, smoking, or corticosteroid therapy).

The primary aim of the study is to investigate the prevalence of these sequelae in the at-risk population of ophthalmologists and orthoptist. Secondary aim are to describe administrative procedures (occupational disease declaration and sick leave), infections characteristics; and risk factors such as a refractive surgery history, the wearing of eyeglasses or contact lenses, smoking, or corticosteroid therapy.

ELIGIBILITY:
Inclusion Criteria:

* Ophtalmologist or orthoptist (interns, graduates and retirees)
* French

Exclusion Criteria:

- Foreign practitionner

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: French Ophtalmologist or orthoptist
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2019-10-21 (Actual); Primary Completion 2022-10 (Estimated); Study Completion 2022-10 (Estimated)

PRIMARY OUTCOMES:
epidemiology characteristics | Day 1
  history of adenovirus keratoconjunctivitis; history of sequels
general characteristics - Sex | Day 1
  general characteristics - Sex
general characteristics - Age range | Day 1
  general characteristics - Age range
general characteristics - Profession | Day 1
  general characteristics - Profession

SECONDARY OUTCOMES:
administrative procedure declaration | Day 1
  occupational disease declaration, sick leave, cessation of surgery and duration
infection characteristics | Day 1
  bilaterality, season, anteriority, sequels, current therapy, professional discomfort
risk factor | Day 1
  refractive surgery history, wearing of eyeglasses or contact lenses, smoking, corticosteroid therapy

CONTACTS AND LOCATIONS:
Locations (1):
- University hospital, Clermont-Ferrand, Clermont-Ferrand, France